CLINICAL TRIAL: NCT01021722
Title: A Modified Surgical Approach to Women With Obstetric Anal Sphincter Tears
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Lund University (Other); Region Skane (Other)
Responsible Party: Pelle Lindqvist, Karolinska University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: sphincter2009
Record Dates: First submitted 2009-11-27; First posted 2009-11-30 (Estimated); Last update posted 2009-11-30 (Estimated); Status verified 2009-11

CONDITIONS: Obstetric Surgical Procedures
Keywords: sphincter; obstetric tears; long-term follow-up

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Modified suture technique (Experimental): Sutured in a modified manner
  Interventions: Procedure: modified suture technique
- Historical sphincter group (No Intervention): The outcome of historical sphincter tears
- Normal primaparous deliveries (No Intervention): Normal deliveries

INTERVENTIONS:
Procedure: modified suture technique — Both internal and external anal sphincter was sutured separately end to end
  Other Names: Historical sphincter tears; Historical normal deliveries
  Arms: Modified suture technique

SUMMARY:
Long-term results after obstetric anal sphincter tears (AST) is poor. The investigators aim to improve the long-term outcome after AST in terms of symptoms of anal incontinence.

A prospective study at, Malmö University Hospital. Twenty-six women with at least grade 3B AST were classified and sutured in a systematic way, including separate suturing of the internal and external sphincter muscles with monofilament absorbable sutures. The principal outcome was a difference in anal incontinence score, based on six questions, between the study group and two control groups (women with prior AST [n = 180] and primiparous women delivered vaginally without AST [n = 100]).

DETAILED DESCRIPTION:
The series was undertaken in advance of a planned prospective randomized controlled study. The study was approved by the Research Ethics Committee of Lund University and informed consent was obtained from all the women involved. Twenty-six women presenting with at least a 3B rupture were recruited by one of the two surgeons (MJ, PL). The modified technique included:

1. Adoption of a structured way of describing the damage according to Fornell an co-workers[7] and recommended by RCOG.[8] Grade 3A: any tear of the ESM < 50% Grade 3B: an ESM tear > 50% Grade 3C: related damage to the ISM Grade 4: related rupture of the anal mucosa
2. The use of monofilament resorbable suture material for all sutures in the mucosa or sphincter muscles. The anal mucosa was sutured with a continuous layer of 3.0 glycomer 631 (Biosyn® ,Tyco Healthcare, Mansfield, MA, USA); the ISM with a continuous layer of 3.0 glycomer 631; and the ESM (both superficial and profound portions) with interrupted end-to-end 2.0 glycomer 631 sutures. The perineal body was usually sutured with 2.0 or 3.0 lactomer (Polysorb®, Tyco Healthcare, Mansfield, MA, USA).
3. Metronidazole 1.5g as a single IV injection and/or Cefuroxime 1.5g IV during the procedure and 6 hours post-operative was usually given as prophylaxis.
4. All women were sutured under either regional anaesthesia (spinal, epidural, or pudendal) or general anaesthesia. Thus, the modified procedure included both a new technique of suturing and the operation was performed by one of the two surgeons involved in the study. Apart from this, all women were treated according to routine departmental practice.

ELIGIBILITY:
Inclusion Criteria:

* Sphincter tear > grad 3B

Exclusion Criteria:

* No

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2002-11; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Differences in anal incontinence score between a study group and two control groups | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pelle G Lindqvist, Principal Investigator — KarolinskaUniversity Hospital
Locations (1):
- UMAS, Malmo, Sweden